CLINICAL TRIAL: NCT07179094
Title: The Effect of a Protective Oral Care Protocol Using Peppermint Oil Mouthwash on Chemotherapy-Induced Nausea, Vomiting, and Loss of Appetite in Patients With Hematologic Malignancies
Brief Title: The Effect of a Protective Oral Care Protocol Using Peppermint Oil Mouthwash
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Şule Güzle (Other)
Responsible Party: Sponsor-Investigator, Şule Güzle, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 125S390
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Neoplasms; Nausea; Vomiting; Anorexia
Keywords: Hematologic Neoplasms; Nausea; Vomiting; Anorexia; Prevention Mouthrinse; peppermint oil
MeSH Terms: conditions — Hematologic Neoplasms; Nausea; Vomiting; Anorexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protective Oral Care Using Peppermint Oil Mouthwash Group (Experimental): The Protective Oral Care Application with Peppermint Oil will begin on the first day of chemotherapy (Day 0) and will continue for the following five days.
  Patients in this group will be instructed to perform oral care with peppermint oil mouthwash three times daily for six consecutive days (Day 0, Day 1, Day 2, Day 3, Day 4, Day 5).
  In addition, patients will be asked to evaluate their throat and oral mucosa immediately before the application, during the application, and 30 minutes after the application using the Allergic Reaction Monitoring Form.
  Peppermint oil mouthwash will be administered at the following times:
  * 07:00-08:00 (morning)
  * 15:00-16:00 (afternoon)
  * 22:00-23:00 (night) At each application, patients will complete the Allergic Reaction Monitoring Form to record local allergic symptoms such as erythema, burning, itching, and sensitivity.
  Interventions: Other: Protective Oral Care Using Peppermint Oil Mouthwash
- Routine Protective Oral Care Group (Active Comparator): Participants in this group will perform oral care according to the routine clinical oral care procedures applied in the oncology clinic. This includes the use of saline solution mouthwash and/or sodium bicarbonate mouthwash. The routine oral care will be carried out on the day of chemotherapy and for the following five days (a total of six consecutive days).
  Interventions: Other: Routine Protective Oral Care

INTERVENTIONS:
Other: Routine Protective Oral Care — In the control group, this group will perform oral care according to the routine clinical oral care procedures applied in the oncology clinic.
  Arms: Routine Protective Oral Care Group
Other: Protective Oral Care Using Peppermint Oil Mouthwash — Patients in the intervention group will perform a mouth rinse three times daily using 1 mL of peppermint oil diluted in 50 mL of water. The first application will be initiated on the day of chemotherapy, and patients will continue the peppermint oil oral care for six consecutive days (Day 0, Day 1, Day 2, Day 3, Day 4, and Day 5). The peppermint oil oral care protocol is scheduled to be administered at 07:00-08:00, 15:00-16:00, and 22:00-23:00, taking into account the routine timing of antiemetic medication administration in the clinic. The detailed description of the oral care protocol is presented below.
  Arms: Protective Oral Care Using Peppermint Oil Mouthwash Group

SUMMARY:
Hematologic malignancies are the fifth most common type of cancer in the world. Patients with hematologic malignancies receive long-term and exhausting treatments such as chemotherapy, radiotherapy, hematopoietic stem cell transplantation and supportive therapies. Chemotherapy-induced nausea and vomiting has a significant impact on the daily lives of patients and causes physiological effects such as anorexia, malnutrition, weight loss, dehydration and electrolyte imbalance. It also has a negative impact on activities of daily living and psychological status, and may lead to poor adherence to chemotherapy regimens, refusal of chemotherapy or discontinuation of treatment. Oral mucosa is one of the areas most affected by the cytotoxic damage of chemotherapy. Disruption of the oral mucosa causes nausea, vomiting and feeding problems. Patients resort to non-drug approaches to manage these problems. It is important that these non-pharmacologic approaches are supported and controlled by reliable and evidence-based studies in order to prevent adverse effects on patient outcomes. In the literature, it has been determined that peppermint oil has antiemetic, antiseptic, anti-inflammatory, analgesic, antiseptic, antioxidant, antiviral, antifungal and spasmolytic effects, protects the integrity of the oral mucosa and has positive effects on nausea-vomiting and anorexia.

In this context, the aim of the study was to investigate the effect of a preventive oral care protocol with peppermint oil mouthwash on chemotherapy-induced nausea, vomiting and appetite in patients with hematologic malignancy.

Research Hypotheses H01: The protective oral care protocol applied with peppermint oil in patients with hematological malignancies has no effect on the development of chemotherapy-induced nausea and vomiting.

H02: The protective oral care protocol applied with peppermint oil in patients with hematological malignancies has no effect on the severity of chemotherapy-induced nausea and vomiting.

H03: The protective oral care protocol applied with peppermint oil in patients with hematological malignancies has no effect on the development of chemotherapy-induced anorexia.

H04: The protective oral care protocol applied with peppermint oil in patients with hematological malignancies has no effect on the severity of chemotherapy-induced anorexia.

Methods: The type of study is a single-blind randomized controlled experimental study. The research will be conducted between September 10, 2025, and April 10, 2026, with patients admitted to the hematology clinic of a university hospital for chemotherapy treatment. The study will be conducted with a total of 72 people who will be randomly assigned to the intervention (n=36) and control groups (n=36) by stratified and block randomization method. Patients who are 18 years of age or older, have hematologic malignancy, with a history of at least one chemotherapy cycle, and scheduled to receive chemotherapy with high or moderate emetogenic risk agents, do not have oral mucositis before chemotherapy, do not have metastasis, are literate and volunteer to participate in the study will be included in the study. Research data will be collected using the "Patient Introduction Form", "Rhodes Nausea-Vomiting and Retching Index", "Oral Assessment Guide", "Appetite Assessment Chart [(Visual Analog Scale (VAS)]", "Peppermint Oil Protective Oral Care Protocol", "Food Intake Record Form", "Allergic Reaction Monitoring Form" and "Patient Monitoring Form and Antiemetic Record Chart". In addition to the routine protective oral care (saline solution mouthwash and/or sodium bicarbonate mouthwash) in the clinic, "Peppermint Oil Protective Oral Care Protocol" will be applied to the intervention group for 6 days from the start of chemotherapy treatment. Patients will receive mouthwash prepared with 1 ml of peppermint oil and 50 ml of prepared drinking water 3 times a day. Patients in the intervention group will be monitored for 6 days by evaluating oral assessment, development of oral mucositis, appetite follow-up and compliance with mouthwash. The development of allergy due to the use of peppermint oil in each mouthwash application will be evaluated. The control group will not receive any oral care intervention by the researcher and will receive routine preventive oral care in the clinic. In the evaluation of the data, descriptive statistics, Chi-square / Fisher's Exact test will be used for the relationship between categorical variables, Mann Whitney U test, Wilcoxon test, Kruskal-Wallis H test will be used for the relationship between continuous variables in groups that do not show normal distribution; one-way analysis of variance / repeated measures analysis of variance, t test for dependent and independent groups will be used in groups with normal distribution. Correlation analysis and regression analysis will be used to examine the relationship between variables.

DETAILED DESCRIPTION:
Background: Hematologic malignancies are a group of neoplasms caused by the uncontrolled proliferation of cells in lymphoid tissue or bone marrow. Hematologic malignancies are considered the fifth most common type of cancer worldwide. Hematologic malignancies are classified differently based on their pathophysiological characteristics, so the treatment method and protocol specific to the type of cancer also varies. Patients face long-term and exhausting treatments such as chemotherapy, radiotherapy, hematopoietic stem cell transplantation, and supportive therapies. Chemotherapy treatment in patients with hematological malignancies causes common symptoms such as pancytopenia, fatigue, oral mucositis, nausea/vomiting, and loss of appetite, depending on the characteristics of the drug. Chemotherapy (CT)-induced nausea and vomiting have a significant impact on patients' daily lives and cause physiological effects such as loss of appetite, malnutrition, weight loss, dehydration, and electrolyte imbalance and physiological effects such as decreased drug absorption or excretion by the kidneys. One of the areas most affected by the cytotoxic damage of chemotherapy is the oral mucosa. Damage to the oral mucosa, nutritional disorders, swallowing disorders, and the development of infections are among the many complications that negatively affect the patient's compliance with treatment. Damage to the oral mucosa associated with chemotherapy, as well as symptoms such as nausea, vomiting, and loss of appetite, can be prevented or reduced through effective nursing interventions and care. In addition to pharmacological methods, non-pharmacological methods are also used in many societies to control nausea, vomiting, and loss of appetite. Herbal products are the most commonly used complementary method by cancer patients to reduce chemotherapy-related side effects. Studies on the effect of herbal products in the management of nausea and vomiting can be found in the literature. A study evaluating the effect of peppermint oil on nausea, vomiting, and loss of appetite in cancer patients has been found. It is stated that medicinal peppermint essential oil may prevent nausea and vomiting due to its spasmolytic and antiseptic effects on the gastric tract and colon. In this context, it is anticipated that this research project, planned as an experimental study, will provide evidence for patient care by determining the effect of peppermint oil oral care on nausea, vomiting, and loss of appetite in patients diagnosed with hematological cancer. The research aims to determine whether a protective peppermint oil oral care protocol reduces the incidence/severity of nausea, vomiting, and loss of appetite in patients with hematological malignancies undergoing chemotherapy.

Methods: The type of study is a single-blind randomized controlled experimental study. The research will be conducted between September 10, 2025, and April 10, 2026, with patients admitted to the hematology clinic of a university hospital for chemotherapy treatment. The study will be conducted with a total of 72 people who will be randomly assigned to the intervention (n=36) and control groups (n=36) by stratified and block randomization method. Patients who are 18 years of age or older, have hematologic malignancy, with a history of at least one chemotherapy cycle, and scheduled to receive chemotherapy with high or moderate emetogenic risk agents, do not have oral mucositis before chemotherapy, do not have metastasis, are literate and volunteer to participate in the study will be included in the study. Individuals will be excluded from the study if they meet any of the following criteria: use of herbal remedies for nausea, vomiting, or anorexia; concurrent radiotherapy with chemotherapy; non-adherence to standard antiemetic therapy according to the chemotherapy preparation regimen and protocol; known allergy to peppermint oil; presence of psychiatric disorders; communication impairments (hearing or speech difficulties); altered level of consciousness; endotracheal intubation; requirement for oral care solutions differing from the clinic's routine procedures (other than saline or sodium bicarbonate); presence of chronic gastrointestinal diseases (including gastritis, gastric/peptic ulcer, ulcerative colitis, Crohn's disease, gastroesophageal reflux, irritable bowel syndrome, cirrhosis, or pancreatitis); migraine; brain metastases; hepatic or renal insufficiency; administration of low-emetogenic chemotherapy; or mucositis, as indicated by an Oral Assessment Guide score reflecting compromised oral health (15-24 points). Research data will be collected using the "Patient Introduction Form", "Rhodes Nausea-Vomiting and Retching Index", "Oral Evaluation Guide", "Appetite Monitoring Chart [(Visual Analog Scale (VAS)]", "Peppermint Oil Protective Oral Care Protocol", "Food Consumption Amount Chart", "Allergic Reaction Monitoring Form" and "Patient Monitoring Form and Antiemetic Record Chart". In addition to the routine preventive oral care (SF and/or sodium bicarbonate mouthwash) in the clinic, "Peppermint Oil Protective Oral Care Protocol" will be applied to the intervention group for 6 days from the start of chemotherapy treatment. Patients will receive mouthwash prepared with 1 ml of peppermint oil and 50 ml of prepared drinking water 3 times a day. Patients in the intervention group will be monitored for 6 days by evaluating oral assessment, development of oral mucositis, appetite follow-up and compliance with mouthwash. The development of allergy due to the use of peppermint oil in each mouthwash application will be evaluated. The control group will not receive any oral care intervention by the researcher and will receive routine preventive oral care in the clinic. In the evaluation of the data, descriptive statistics, Chi-square / Fisher's Exact test will be used for the relationship between categorical variables, Mann Whitney U test, Wilcoxon test, Kruskal-Wallis H test will be used for the relationship between continuous variables in groups that do not show normal distribution; one-way analysis of variance / repeated measures analysis of variance, t test for dependent and independent groups will be used in groups with normal distribution. Correlation analysis and regression analysis will be used to examine the relationship between variables.

The detailed description of the oral care protocol is presented below. Peppermint Oil Protective Oral Care Protocol

1. Materials

   * 1 ml peppermint oil
   * 1 disposable paper cup
   * 1 wooden stir stick
   * 50 ml bottled water or boiled and cooled tap water
2. Preparation of Peppermint Oil Mouthwash

   * Wash and dry hands thoroughly.
   * Pour 50 ml of bottled water or boiled and cooled tap water into the paper cup.
   * Add 1 ml of peppermint oil (kept at room temperature) into the cup.
   * Mix the water and peppermint oil using the wooden stir stick.
3. Application of Peppermint Oil Mouthwash

   * If lying in bed, sit upright before the procedure.
   * Take approximately 5 ml of the prepared solution into the mouth and gargle.
   * Gargle for about 30 seconds, then spit out the solution.
   * Do not swallow the solution.
   * If any discomfort occurs in the oral cavity, stop the procedure immediately and inform the researcher.
   * After completing the procedure, discard the used materials and wash your hands.
4. Recording of Mouthwash Application

   • Document the procedure in the Patient Monitoring Form.
5. Precautions

   * Perform peppermint oil mouthwash three times daily at the following times:

     * 07:00-08:00
     * 15:00-16:00
     * 22:00-23:00
   * Mouthwash use should begin concurrently with chemotherapy treatment.
   * Avoid drinking liquids or consuming food, and refrain from rinsing the mouth for at least 30 minutes after using the mouthwash.
   * Continue routine clinical oral care practices in addition to peppermint oil mouthwash.
   * Store peppermint oil at room temperature in a dark place away from direct light.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of hematologic malignancy
* History of at least one chemotherapy cycle
* Scheduled to receive chemotherapy with high or moderate emetogenic risk agents
* No oral mucositis before chemotherapy
* No metastasis
* Literate (able to read and write)
* Volunteer to participate in the study

Exclusion Criteria:

* Use of herbal remedies for nausea, vomiting, or anorexia
* Concurrent radiotherapy with chemotherapy
* Non-adherence to standard antiemetic therapy according to the chemotherapy preparation regimen and protocol (e.g., use of antiemetics other than granisetron or metoclopramide)
* Known allergy to peppermint oil
* Psychiatric disorders
* Communication impairments (hearing or speech difficulties)
* Altered level of consciousness
* Endotracheal intubation
* Requirement for oral care solutions other than the clinic's routine procedures (saline or sodium bicarbonate)
* Chronic gastrointestinal diseases (gastritis, gastric/peptic ulcer, ulcerative colitis, Crohn's disease, gastroesophageal reflux, irritable bowel syndrome, cirrhosis, or pancreatitis)
* Migraine
* Brain metastases
* Hepatic or renal insufficiency
* Administration of low-emetogenic chemotherapy
* Mucositis (Oral Assessment Guide score: 15-24 points)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Nausea-Vomiting-Retching Symptoms | 7 months
  The nausea, vomiting, and retching symptoms that may develop due to chemotherapy will be assessed using the Rhodes Index of Nausea, Vomiting, and Retching (RINVR).
  The scale consists of eight items measuring the frequency, duration, and severity of symptoms. In scoring, each response ranges from 0 (no distress) to 4 (maximum distress). The patient's experiences across all eight items are summed, with a maximum possible score of 32, indicating the most severe symptom burden. The index comprises three sub-dimensions: symptom experience, symptom occurrence, and symptom distress.
  Assessments will begin one day prior to chemotherapy and will continue on the day of chemotherapy and for five consecutive days thereafter.
Oral Health Status | 7 months
  The oral mucosal conditions of participants will be evaluated using the Oral Assessment Guide (OAG). This guide assesses dentures, teeth, gums, mucous membranes, saliva, tongue, lips, swallowing, and voice. Each item is scored from 1 to 3, and total scores are obtained by summation, ranging between 8 and 24. Lower scores indicate better oral health, while higher scores reflect deterioration.
  According to the OAG:
  * 8-14 points: At risk for oral health deterioration
  * 15-24 points: Presence of oral health deterioration Evaluations will begin one day prior to chemotherapy and will be conducted on the chemotherapy day and for five consecutive days thereafter.
Anorexia Symptom | 7 months
  Participants' anorexia symptoms will be assessed using the Appetite Assessment Chart [Visual Analog Scale (VAS)]. The chart consists of a 100 millimeters horizontal line, and scores are determined by measuring the distance (in mm) between the left anchor and the point marked by the patient.
  * Left anchor (0): "My appetite is very good"
  * Right anchor (10): "I have no appetite at all" Scores range from 0 to 10, with higher scores indicating greater severity of anorexia symptoms. Participants will be asked to make one marking per 24-hour period to reflect their appetite status. Assessments will start one day prior to chemotherapy and will continue on the day of chemotherapy and for five consecutive days thereafter.

SECONDARY OUTCOMES:
Food Intake Status | 7 months
  Participants' food intake at meals will be recorded using the Food Intake Record Form. This tool will be used to evaluate how anorexia symptoms develop and their impact on nutritional intake. The form covers breakfast, lunch, dinner, and snacks, with consumption at each meal rated in percentage categories (0%, 25%, 50%, 75%, 100%). Daily intake will be calculated by summing the percentages across meals. Records will start one day prior to chemotherapy and continue on the chemotherapy day and for five consecutive days thereafter.
Adherence and Monitoring of Peppermint Oil-Based Protective Oral Care | 7 months
  A Patient Monitoring Form will be created separately for the intervention and control groups. The form will include: RINVR scores, oral care assessment score, food intake records, appetite chart scores, oral care adherence, and allergic reaction follow-up. The form also includes information on the dates and time range (7 days / 10:00 PM-11:00 PM) of peppermint oil mouthwash application and protective oral care, as well as the name and dose of the antiemetic medication. Patients will be asked to document the times at which they perform oral care and complete the scales.
  Participants in the intervention group will perform peppermint mouthwash three times daily (morning, noon, evening) as part of the Peppermint Oil Protective Oral Care Protocol. Compliance will be documented in the Patient Monitoring Form. Gargling will begin on the day of chemotherapy and continue for five days thereafter.
Monitoring of Allergic Reactions | 7 months
  The Allergic Reaction Monitoring Form will be used to examine adverse reactions associated with peppermint oil oral care. Participants in the intervention group will be evaluated with this form prior to, during, and 30 minutes after gargling. Local allergic symptoms such as mucosal erythema, burning, itching, and sensitivity will be recorded. Monitoring will start on the chemotherapy day and continue for five consecutive days.
Anthropometric Measurements | 7 months
  Biomarkers that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Participants' height (m) and weight (kg) will be measured and used to calculate Body Mass Index (BMI, kg/m²). Height and weight are combined to report a single BMI value. Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.
  • Unit of Measure: kg/m²
Biochemical Findings - mg/dL | 7 months
  Biomarkers that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Routine biochemical tests performed in the clinic will be retrieved from hospital records, measured in mg/dL, including:
  * Total cholesterol
  * Creatinine
  * Bilirubin
    * Unit of Measure: mg/dL Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.
Biochemical Findings - g/dL | 7 months
  Biomarkers that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Routine biochemical tests performed in the clinic will be retrieved from hospital records, measured in g/dL, including:
  * Albumin
  * Total protein
    * Unit of Measure: g/dL
    * Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.
Biochemical Findings - mEq/L | 7 months
  Biomarker that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Routine biochemical test performed in the clinic will be retrieved from hospital records, measured in mEq/L, including:
  o Sodium Unit of Measure: mEq/L Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.
Biochemical Findings - µg/dL | 7 months
  Biomarker that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Routine biochemical test performed in the clinic will be retrieved from hospital records, measured in µg/dL, including:
  o Iron
  * Unit of Measure: µg/dL
  * Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.
Biochemical Findings - count/µL | 7 months
  Biomarkers that may be affected by nausea, vomiting, and anorexia symptoms-and thus influence nutritional status and patient outcomes-will be monitored. Routine biochemical tests performed in the clinic will be retrieved from hospital records, measured in count/µL, including:
  o Neutrophil
  * Unit of Measure: count/µL
  * Data will be collected one day prior to chemotherapy and on the fifth day of chemotherapy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tipton JM, McDaniel RW, Barbour L, Johnston MP, Kayne M, LeRoy P, Ripple ML. Putting evidence into practice: evidence-based interventions to prevent, manage, and treat chemotherapy-induced nausea and vomiting. Clin J Oncol Nurs. 2007 Feb;11(1):69-78. doi: 10.1188/07.CJON.69-78. PMID 17441398
- [Background] Khaddour K, Hana CK, Mewawalla P. Hematopoietic Stem Cell Transplantation. 2023 May 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536951/ PMID 30725636
- [Background] Kennedy SKF, Goodall S, Lee SF, DeAngelis C, Jocko A, Charbonneau F, Wang K, Pasetka M, Ko YJ, Wong HCY, Chan AW, Rajeswaran T, Gojsevic M, Chow E, Gralla RJ, Ng TL, Jerzak KJ. 2020 ASCO, 2023 NCCN, 2023 MASCC/ESMO, and 2019 CCO: a comparison of antiemetic guidelines for the treatment of chemotherapy-induced nausea and vomiting in cancer patients. Support Care Cancer. 2024 Apr 10;32(5):280. doi: 10.1007/s00520-024-08462-x. PMID 38594320
- [Background] Evans A, Malvar J, Garretson C, Pedroja Kolovos E, Baron Nelson M. The Use of Aromatherapy to Reduce Chemotherapy-Induced Nausea in Children With Cancer: A Randomized, Double-Blind, Placebo-Controlled Trial. J Pediatr Oncol Nurs. 2018 Nov/Dec;35(6):392-398. doi: 10.1177/1043454218782133. Epub 2018 Jun 27. PMID 29947285
- [Background] Tavakoli Ardakani M, Ghassemi S, Mehdizadeh M, Mojab F, Salamzadeh J, Ghassemi S, Hajifathali A. Evaluating the effect of Matricaria recutita and Mentha piperita herbal mouthwash on management of oral mucositis in patients undergoing hematopoietic stem cell transplantation: A randomized, double blind, placebo controlled clinical trial. Complement Ther Med. 2016 Dec;29:29-34. doi: 10.1016/j.ctim.2016.08.001. Epub 2016 Aug 30. PMID 27912953
- [Background] Jafarimanesh H, Akbari M, Hoseinian R, Zarei M, Harorani M. The Effect of Peppermint (Mentha piperita) Extract on the Severity of Nausea, Vomiting and Anorexia in Patients with Breast Cancer Undergoing Chemotherapy: A Randomized Controlled Trial. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420967084. doi: 10.1177/1534735420967084. PMID 33118401
- See also: Randomization — https://randomizer.org/